CLINICAL TRIAL: NCT04367857
Title: SARS-CoV-2 Seroprevalence Among Healthcare Workers: ARMOR Study Demonstration Project
Brief Title: ARMOR Study: COVID-19 Seroprevalence Among Healthcare Workers
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAS9998
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Covid-19; Coronavirus Infection; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prior Positive polymerase chain reaction (PCR) and Recovered: Prior Positive PCR result, fully recovered, back at work and symptom free for greater than or equal than 14 days.
  Interventions: Other: COVID-19 Serology; Behavioral: Health Care Worker Survey
- Never tested, history of COVID-19 Symptoms and Recovered: Never tested and history of COVID-19 symptoms and symptom-free for more than 14 days
  Interventions: Other: COVID-19 Serology; Behavioral: Health Care Worker Survey
- Never tested and current COVID-19 Symptoms: Never tested and current COVID-19 Symptoms (e.g. referred by a provider or clinic)
  Interventions: Other: COVID-19 Serology; Behavioral: Health Care Worker Survey
- Never tested and asymptomatic: Never tested and asymptomatic for COVID-19 symptoms, including asymptomatic health care worker
  Interventions: Other: COVID-19 Serology; Behavioral: Health Care Worker Survey

INTERVENTIONS:
Other: COVID-19 Serology — Quantitate Serology enzyme-linked immunosorbent assay (ELISA) for COVID-19
Behavioral: Health Care Worker Survey — The purpose of this survey is to assess how healthcare workers are experiencing and coping with the COVID-19 crisis.

SUMMARY:
The novel coronavirus (SARS-CoV-2) has spread all around the world and testing has posed a challenge globally. Health care providers are highly exposed and are an important group to test. On top of these concerns, health care workers are also stressed by the needs on responders in the COVID-19 crisis. The investigators will look at different ways to measure how common COVID-19 is among health care workers, how common is the presence of antibodies by serological tests (also known as serostatus). The investigators will describe health worker mental and emotional well-being and their coping strategies in their institutional settings. Lastly, the investigators will describe how knowing serostatus can affect individuals' mental and emotional well-being and how to cope in the midst of the COVID-19 response. This will help to how to better test and help healthcare workers in the COVID-19 pandemic and prepare for possible future outbreaks.

DETAILED DESCRIPTION:
The rapid spread of the novel coronavirus SARS-CoV-2 has resulted in pandemic levels and a global challenge in diagnosing infection. Diagnosing infection, defining recovery and immunity has been challenging. Health care providers in particular are very interested in knowing their status as they are highly exposed, and if infectious, can potentially transmit infection nosocomially (in the healthcare workplace setting) and to their household. In addition to understanding their exposure risk, infectious period, and immunity status, health care workers are reporting high levels of psychosocial distress including anxiety and burnout. The investigators aim to assess the baseline and cumulative seroprevalence of SARS-CoV-2 among health care workers using both quantitative and qualitative serological assays; describe psychosocial well-being and coping strategies among health workers in their institutional settings and describe how knowledge of one's serostatus affect psychosocial well-being, and coping strategies. Findings from this study will inform; 1) use of serological assays and testing algorithms, and 2) approaches to manage psychosocial stress for healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* NewYork-Presbyterian (NYP) healthcare personnel employee or affiliate
* Understands and reads English

Exclusion Criteria:

* Younger than 18 years of age
* Mentally and/or physically unable to complete study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employee of NewYork-Presbyterian Hospital and its affiliates
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion seropositive | Up to 12 months after collection visit
  Percentage of health care workers with positive serological markers to describe patterns in exposure, re-infection, clinical symptom, serological responses among health care workers based on their baseline serological status over a one year period.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Sobieszczyk, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- NewYork-Presbyterian Hosptial/Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided